CLINICAL TRIAL: NCT04531540
Title: HT201321- Repeated Insult Patch Test With Modified Challenge
Brief Title: Study to Determine Skin Irritation and/or Sensitization Potential of an Antifungal Cream Containing Trolamine (Repeated Insult Patch Test)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18156
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — butenafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Repeated Insult Patch Test (Experimental): During the Induction Phase, participants received 0.2 g Butenafine HCl 1% covered by an occlusive patch on the upper back skin test site three times a week for a total of 9 applications. Prior to each patch application and after the last patch removal, the test sites were evaluated for gross changes according to the Erythemal Scoring Scale and if necessary the Additional Scoring system. After 14 days of Rest Phase, on the first day of Challenge Phase, participants received same procedure on original Induction Phase test site and on a virgin test site. The patches were removed and the sites scored 48 hours after application and scored again at 96 hours after application. The test sites were evaluated using the Induction Phase scoring system.
  Interventions: Drug: Butenafine HCl 1% (BAY1896425)

INTERVENTIONS:
Drug: Butenafine HCl 1% (BAY1896425) — Approximately 0.2 g of cream containing butenafine HCl 1% were applied to the upper back skin.
  Other Names: Antifungal Cream V61-044 containing Trolamine

SUMMARY:
In this study researcher want to learn more about possible skin reactions such after repeated application of an antifungal cream containing Trolamine. They are especially interested in skin irritations or allergic skin reactions. The study plans to enroll about 225 female or male participants with the age 18 - 79 years. The antifungal test cream will be applied on the back between the shoulder blades of the participants and covered by a special dressing patch. This will be repeated 3 times a week for the first 3 weeks of this study applying the cream on the same area of the back. At each visit the skin will be investigated for redness, dryness and other reactions. After a rest period of two weeks the test cream will be applied on the same skin area as before and on a second new skin area nearby. After 2 and 4 days the two skin areas will again be investigated for redness, dryness and other reactions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been aged 18 to 79 years, inclusive;
* Female subjects must have produced a negative urine pregnancy test prior to the initiation and also at the completion of the trial;
* Subjects must have been capable of understanding and following directions.

Exclusion Criteria:

* Subjects who were in ill health or taking medication, other than birth control, which could influence the purpose, integrity or outcome of the trial;
* Subjects who had any visible skin disease that might be confused with a skin reaction to the test material;
* Subjects who were participating in another clinical trial at this facility or any other facility;
* Subjects who used topical or systemic steroids or antihistamines for at least 7 days prior to trial initiation and during the duration of the trial;
* Subjects who had a history of adverse reactions to adhesive tape, cosmetics, OTC drugs or other personal care products;
* Subjects judged by the PI to be inappropriate for the trial;
* Female subjects who were pregnant as evidenced by a urine pregnancy test, planning to become pregnant, or nursing during the course of the trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2013-10-18 (Actual); Study Completion 2013-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at single center in the US, between 9 SEP 2013 (first subject first visit) and 18 OCT 2013 (last subject last visit).
Pre-assignment Details: A total of 225 subjects were enrolled in the study and 222 received study treatment.
Period: Overall Study
Arm/Group | Repeated Insult Patch Test
Started | 225
Treated | 222
Completed | 216
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 4
Not completed — Found to be Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Repeated Insult Patch Test
Number analyzed (Participants) | 225
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 66
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 154
  Hispanic | 38
  Caucasian/Hispanic | 3
  African American | 23
  Caucasian/African American | 1
  Caucasian/American Indian | 1
  American Indian | 1
  Asian | 3
  Not Available | 1

OUTCOME MEASURES:

1. Primary Outcome: Irritation Response Evaluation According to Erythema Scoring Scale During Induction Phase - All Enrolled Subjects
Description: Prior to each patch application and after the last patch removal, the test sites were evaluated for gross changes according to the Erythema Scoring Scale: score 0=No visible erythema; score 0.5=Slight, barely perceptible erythema; score 1=Mild erythema; score 2=Moderate erythema; score 3=Marked erythema; score 4=Severe erythema.
Time Frame: After 4 weeks
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Repeated Insult Patch Test
Number analyzed (Participants) | 225
Number analyzed (Test site) | 2184
Test site
  score=0 | 2182
  score=0.5 | 2

2. Primary Outcome: Allergic Reaction Evaluation According to Erythema Scoring Scale During Challenge Phase - All Enrolled Subjects
Description: as for outcome 1
Time Frame: After 6 weeks
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Repeated Insult Patch Test
Number analyzed (Participants) | 225
Number analyzed (Test site) | 1296
Test site
  score=0 | 1296
  score=0.5 | 0

3. Primary Outcome: Irritation Response Evaluation According to Erythema Scoring Scale During Induction Phase - All Evaluable Subjects
Description: as for outcome 1
Time Frame: After 4 weeks
Population: Subjects who received treatment and completed the trial and had evaluable data
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Repeated Insult Patch Test
Number analyzed (Participants) | 216
Number analyzed (Test site) | 2160
Test site
  score=0 | 2158
  score=0.5 | 2

4. Primary Outcome: Allergic Reaction Evaluation According to Erythema Scoring Scale During Challenge Phase - All Evaluable Subjects
Description: as for outcome 1
Time Frame: After 6 weeks
Population: Subjects who received treatment and completed the trial and had evaluable data
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Repeated Insult Patch Test
Number analyzed (Participants) | 216
Number analyzed (Test site) | 1296
Test site
  score=0 | 1296
  score=0.5 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Repeated Insult Patch Test
Serious Adverse Events (participants affected / at risk) | 0/225
Other Adverse Events (participants affected / at risk) | 6/225
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Repeated Insult Patch Test (N=225)
Headache (Nervous system disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 1
Other - Irritation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No information based on the conduct of the study (incl. protocol, data resulting from the study, or the fact that the study was being conducted) will be released without prior written consent of the sponsor unless the requirement is superseded by State or Federal law.